CLINICAL TRIAL: NCT04390295
Title: Clinical Trial to Evaluate the Efficacy and Safety of SHR3824 Combined With Metformin in Metformin Monotherapy Poorly Glycemic Controlled Chinese Type 2 Diabetic Patients
Brief Title: Efficacy and Safety of SHR3824 in Combination With Metformin in Subjects With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR3824-302
Record Dates: First submitted 2018-09-18; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — henagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR3824+Metformin, Placebo+Metformin (Experimental): once daily for SHR3824 and placebo, three times daily for metformin, 24 weeks
  Interventions: Drug: Placebo
- SHR3824 5 mg+Metformin (Experimental): once daily for SHR3824, three times daily for metformin, 52 weeks
  Interventions: Drug: SHR3824; Drug: metformin
- SHR3824 10 mg+Metformin (Experimental): once daily for SHR3824, three times daily for metformin, 52 weeks
  Interventions: Drug: SHR3824; Drug: metformin

INTERVENTIONS:
Drug: Placebo — Once daily, 24 weeks
  Arms: SHR3824+Metformin, Placebo+Metformin
Drug: SHR3824 — Once daily, 52 weeks
  Arms: SHR3824 10 mg+Metformin; SHR3824 5 mg+Metformin
Drug: metformin — Three times daily, 52 weeks
  Arms: SHR3824 10 mg+Metformin; SHR3824 5 mg+Metformin

SUMMARY:
The purpose of this study is to obtain information on efficacy and safety of SHR3824 with metformin over 24 weeks and 52 weeks in metformin monotherapy poorly glycemic controlled chinese Type 2 Diabetes. Efficacy and safety will be evaluated by comparing the effect of SHR3824 with metformin to placebo with metformin when given in oral doses.

DETAILED DESCRIPTION:
A phase III clinical study on efficacy and safety of SHR3824 combined with metformin for type 2 diabetes with poor glucose control in metformin monotherapy (multicenter, randomized, double-blind, placebo-parallel control). The 450 subjects received at least eight weeks of metformin monotherapy at a steady dose of 1500 mg or more before screening.

Evaluation of efficacy: compared with the group of placebo combined with metformin, HbA1c, fasting plasma glucose, postprandial plasma glucose, fasting body weight and blood pressure changes in the SHR3824 with metformin group

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of type 2 diabetes mellitus;
* Patients with type 2 diabetes mellitus treated with metformin monotherapy for ≥ 8 weeks and poor glycemic control, metformin dose stabilized ≥1500mg / day;
* FPG<=15mmol/L;
* Hemoglobin A1c levels >=7.0% and <=10.5%;
* Body mass index (BMI) 19 to 35 kg/m2;

Exclusion Criteria:

* Type I diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes mellitus (acromegaly, Cushing's syndrome, etc.);
* Past or current history of severe diabetic complications (proliferative diabetic retinopathy, stage III or later stage overt nephropathy, diabetic ketoacidosis, or serious diabetic neuropathy);
* Systolic blood pressure of ≥160 mmHg or diastolic blood pressure of ≥100 mmHg on the start or end day of the run-in period;
* History of myocardial infarction, unstable angina, or cerebrovascular disorder within 6 months before the start of the run-in period;
* Past or current history of malignant tumor;
* Past or current history of drug hypersensitivity such as shock and anaphylactoid symptoms;
* Pregnant women, lactating mothers, or women of childbearing potential;
* Any condition that subjects are assessed to be ineligible by the investigator (sub investigator).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Adjusted Mean Change in HbA1c Levels | Baseline to Week 24
  Compared with the placebo with metformin group, mean change in HbA1c Levels in SHR3824 with metformin group

SECONDARY OUTCOMES:
Adjusted Mean Change in Fasting Plasma Glucose | Baseline to Week 24
  Compared with the placebo with metformin group, mean change in Fasting Plasma Glucose Levels in SHR3824 with metformin group
The number of volunteers with adverse events as a measurement of safety | Baseline to Week 52
  Compared with the placebo with metformin group, the incidence of adverse events in SHR3824 with metformin group

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital of Sun Yat - sen University, Guangzhou, Guangdong, China